CLINICAL TRIAL: NCT00983684
Title: TARGIT: A Randomised Controlled Trial to Compare Targeted Intra-operative Radiotherapy With Conventional Post-operative Radiotherapy After Conservative Breast Surgery for Women With Early Stage Breast Cancer
Brief Title: Comparison of Intra-operative Radiotherapy With Post-operative Radiotherapy for Women With Early Breast Cancer
Acronym: TARGIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN 34086741; ISRCTN 34086741; MREC No. 99/0307; UKCRN ID 7265
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Invasive Breast Cancer; Breast Cancer
Keywords: Neoplasms by Site; Breast Neoplasms; Breast Diseases; Breast Cancer; Cancer of Breast; Cancer of the Breast; Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Neoplasms by Site; Breast Diseases; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-operative radiotherapy (Experimental): A single fraction of radiotherapy given intra-operatively and targeted to the tissues at the highest risk of local recurrence.
  Interventions: Device: Intrabeam
- Post-operative radiotherapy (Active Comparator): Standard post-operative radiotherapy.
  Interventions: Radiation: Post-operative radiotherapy

INTERVENTIONS:
Device: Intrabeam — A dose of 20 Gy at the surface of the applicator or 6 Gy at 1cm (in water) is prescribed by the radiation oncologist and delivered to the breast tissue. This takes approximately 30 minutes, depending on the size of the applicator.
  Other Names: IORT, targeted intra-operative radiotherapy, TARGIT
  Arms: Intra-operative radiotherapy
Radiation: Post-operative radiotherapy — All patients randomised to receive conventional radiotherapy within this trial should be treated in accordance with a pre-specified policy. Dosage should only be applied to the breast; axillary, supra-clavicular and internal mammary nodes should not generally be irradiated by discrete fields.
  Other Names: EBRT
  Arms: Post-operative radiotherapy

SUMMARY:
The purpose of this study is to evaluate whether a single fraction of radiotherapy given intra-operatively and targeted to the tissues at the highest risk of local recurrence is equivalent to standard post-operative external beam radiotherapy after breast conserving surgery in women with early stage breast cancer in terms of local relapse within the treated breast.

DETAILED DESCRIPTION:
TARGIT is an international randomised clinical trial designed to test the hypothesis that the strategy of delivering a single dose of targeted intraoperative radiotherapy (IORT) in patients eligible for breast conserving therapy (with the addition of whole breast radiotherapy in those patients at high risk of recurrence elsewhere in the breast [e.g. lobular carcinomas and extensive intraductal component]) is equivalent to a conventional course of post-operative external beam radiotherapy (EBRT). The primary endpoints are local and loco-regional recurrence rates. It is a pragmatic trial in which each participating centre has the option to define more restrictive entry criteria than in the core protocol. Only centres with access to the Intrabeam® (Carl Zeiss) enter patients into the trial. Eligible patients are those with tumours of good prognosis suitable for breast conserving surgery. After giving consent patients are randomised to either IORT or to EBRT. They may receive any other adjuvant treatments as deemed necessary, except for neoadjuvant therapy. The protocol requires that patients be followed at six monthly intervals for five years and then annually.

ELIGIBILITY:
Inclusion criteria

* Age 45 years or older
* Operable invasive breast cancer (T1 and small T2, N0-1, M0) confirmed by cytological or histological examination
* Suitable for breast conserving surgery
* Previously diagnosed and treated contralateral breast cancer may be entered but will be randomised to a separate stratum.
* Available for regular follow-up for at least ten years.

Note: Individual centres may wish to restrict entry to a more exactly defined subset of patients, in which case, only patients with these characteristics may be entered by that particular centre. For example, centres may decide at outset to recruit only women over 50 or even over 65 years of age. Such policies must be pre-defined in writing and approved by the International Steering Committee.

Exclusion criteria

* More than one obvious cancer in the same breast as diagnosed by clinical examination, mammography or ultrasonography.
* Bilateral breast cancer at the time of diagnosis.
* Ipsilateral breast had a previous cancer and/or irradiation.
* Patients known to have BRCA2 gene mutations, but testing for gene mutations is not required
* Lobular cancer or Extensive intraductal Component (EIC =>25% of the tumour is intraductal) on core biopsy or initial pathology (if performed)
* Patients undergoing primary medical treatment (hormones or chemotherapy) as initial treatment with neoadjuvant intent of reducing tumour size should be excluded; those given short duration (up to 4 weeks) systemic therapy can be included.
* Patients presenting with gross nodal disease, considered to be clinically malignant or proven cytologically or by scanning. In general, 4 or more positive nodes or extranodal spread are not suitable for Targit alone and should receive EBRT as well. However, individual centres may decide that anything more than micrometastasis should receive EBRT.
* Patients with any severe concomitant disease that may limit their life expectancy.
* Previous history of malignant disease does not preclude entry if the expectation of relapse-free survival at 10 years is 90% or greater.
* Any factor included as exclusion criterion in the local centre's Treatment Policy. This is particularly relevant to patients entered into the post pathology stratum.
* No more than 30 days can have elapsed between last breast cancer surgery (not axillary) and entry into the trial for patients in the post-pathology stratification.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3451 (Actual)
Dates: Start 2000-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Local relapse within the treated breast. | 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96, 108, 120 months

SECONDARY OUTCOMES:
Site of relapse within the breast | 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96, 108, 120 months
Relapse-free survival and overall survival | 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96, 108, 120 months
Local toxicity/morbidity | 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96, 108, 120 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Tobias, MD FRCP FRCR, Principal Investigator — University College London Hospitals
Locations (1):
- Clinical Trials Group, London, United Kingdom

REFERENCES:
- [Result] Vaidya JS, Joseph DJ, Tobias JS, Bulsara M, Wenz F, Saunders C, Alvarado M, Flyger HL, Massarut S, Eiermann W, Keshtgar M, Dewar J, Kraus-Tiefenbacher U, Sutterlin M, Esserman L, Holtveg HM, Roncadin M, Pigorsch S, Metaxas M, Falzon M, Matthews A, Corica T, Williams NR, Baum M. Targeted intraoperative radiotherapy versus whole breast radiotherapy for breast cancer (TARGIT-A trial): an international, prospective, randomised, non-inferiority phase 3 trial. Lancet. 2010 Jul 10;376(9735):91-102. doi: 10.1016/S0140-6736(10)60837-9. PMID 20570343
- [Result] Vaidya JS, Wenz F, Bulsara M, Tobias JS, Joseph DJ, Keshtgar M, Flyger HL, Massarut S, Alvarado M, Saunders C, Eiermann W, Metaxas M, Sperk E, Sutterlin M, Brown D, Esserman L, Roncadin M, Thompson A, Dewar JA, Holtveg HM, Pigorsch S, Falzon M, Harris E, Matthews A, Brew-Graves C, Potyka I, Corica T, Williams NR, Baum M; TARGIT trialists' group. Risk-adapted targeted intraoperative radiotherapy versus whole-breast radiotherapy for breast cancer: 5-year results for local control and overall survival from the TARGIT-A randomised trial. Lancet. 2014 Feb 15;383(9917):603-13. doi: 10.1016/S0140-6736(13)61950-9. Epub 2013 Nov 11. PMID 24224997
- [Derived] Vaidya JS, Bulsara M, Baum M, Wenz F, Massarut S, Pigorsch S, Alvarado M, Douek M, Saunders C, Flyger H, Eiermann W, Brew-Graves C, Williams NR, Potyka I, Roberts N, Bernstein M, Brown D, Sperk E, Laws S, Sutterlin M, Corica T, Lundgren S, Holmes D, Vinante L, Bozza F, Pazos M, Blanc-Onfroy ML, Gruber G, Polkowski W, Dedes KJ, Niewald M, Blohmer J, McReady D, Hoefer R, Kelemen P, Petralia G, Falzon M, Joseph D, Tobias JS. New clinical and biological insights from the international TARGIT-A randomised trial of targeted intraoperative radiotherapy during lumpectomy for breast cancer. Br J Cancer. 2021 Aug;125(3):380-389. doi: 10.1038/s41416-021-01440-8. Epub 2021 May 25. PMID 34035435
- [Derived] Vaidya JS, Bulsara M, Baum M, Wenz F, Massarut S, Pigorsch S, Alvarado M, Douek M, Saunders C, Flyger HL, Eiermann W, Brew-Graves C, Williams NR, Potyka I, Roberts N, Bernstein M, Brown D, Sperk E, Laws S, Sutterlin M, Corica T, Lundgren S, Holmes D, Vinante L, Bozza F, Pazos M, Le Blanc-Onfroy M, Gruber G, Polkowski W, Dedes KJ, Niewald M, Blohmer J, McCready D, Hoefer R, Kelemen P, Petralia G, Falzon M, Joseph DJ, Tobias JS. Long term survival and local control outcomes from single dose targeted intraoperative radiotherapy during lumpectomy (TARGIT-IORT) for early breast cancer: TARGIT-A randomised clinical trial. BMJ. 2020 Aug 19;370:m2836. doi: 10.1136/bmj.m2836. PMID 32816842
- [Derived] Vaidya JS, Bulsara M, Saunders C, Flyger H, Tobias JS, Corica T, Massarut S, Wenz F, Pigorsch S, Alvarado M, Douek M, Eiermann W, Brew-Graves C, Williams N, Potyka I, Roberts N, Bernstein M, Brown D, Sperk E, Laws S, Sutterlin M, Lundgren S, Holmes D, Vinante L, Bozza F, Pazos M, Le Blanc-Onfroy M, Gruber G, Polkowski W, Dedes KJ, Niewald M, Blohmer J, McCready D, Hoefer R, Kelemen P, Petralia G, Falzon M, Baum M, Joseph D. Effect of Delayed Targeted Intraoperative Radiotherapy vs Whole-Breast Radiotherapy on Local Recurrence and Survival: Long-term Results From the TARGIT-A Randomized Clinical Trial in Early Breast Cancer. JAMA Oncol. 2020 Jul 1;6(7):e200249. doi: 10.1001/jamaoncol.2020.0249. Epub 2020 Jul 9. PMID 32239210
- [Derived] Vaidya JS, Wenz F, Bulsara M, Tobias JS, Joseph DJ, Saunders C, Brew-Graves C, Potyka I, Morris S, Vaidya HJ, Williams NR, Baum M. An international randomised controlled trial to compare TARGeted Intraoperative radioTherapy (TARGIT) with conventional postoperative radiotherapy after breast-conserving surgery for women with early-stage breast cancer (the TARGIT-A trial). Health Technol Assess. 2016 Sep;20(73):1-188. doi: 10.3310/hta20730. PMID 27689969